CLINICAL TRIAL: NCT03176459
Title: A Multicenter, Randomized, Double-blind, Active-controlled Study to Evaluate the Safety and Efficacy of EXPAREL When Administered Via Infiltration Into the Transversus Abdominis Plane (TAP) Versus Bupivacaine Alone in Subjects Undergoing Elective Cesarean Section
Brief Title: Evaluate the Safety and Efficacy of EXPAREL When Administered Via Infiltration Into the TAP vs. Bupivacaine Alone in Subjects Undergoing Elective C-Sections
Acronym: C-Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 402-C-411
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: C-Section; Pain Management
Keywords: bupivacaine; exparel; analgesic; TAP Block
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double-Blind Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPAREL+bupivacaine TAP infiltration (Experimental): Receive a single 20-mL dose of EXPAREL 266 mg expanded in volume with 20 mL normal saline plus 20 mL 0.25% bupivacaine for a total volume of 60 mL.
  Interventions: Drug: Exparel + Bupivacaine
- Active bupivacaine TAP infiltration (Active Comparator): Receive 20 mL 0.25% bupivacaine expanded in volume with 40 mL normal saline for a total volume of 60 mL
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Exparel + Bupivacaine — EXPAREL is a local analgesic that utilizes bupivacaine in combination with the proven product delivery platform, DepoFoam®.
  Arms: EXPAREL+bupivacaine TAP infiltration
Drug: Bupivacaine — Bupivacaine Hydrochloride is indicated for the production of local or regional anesthesia or analgesia for surgery, dental and oral surgery procedures, diagnostic and therapeutic procedures, and for obstetrical procedures.
  Arms: Active bupivacaine TAP infiltration

SUMMARY:
Primary objective: The primary objective of this study is to compare total opioid consumption through 72 hours following EXPAREL+bupivacaine HCl infiltration into the transversus abdominis plane (TAP) after spinal anesthesia to active bupivacaine HCl TAP infiltration after spinal anesthesia in subjects undergoing an elective cesarean section (C-section).

Secondary objective: The secondary objectives are to assess efficacy and safety parameters and patient satisfaction.

DETAILED DESCRIPTION:
This is a Phase-4, multicenter, randomized, double-blind, active-controlled study planned in approximately 152 adult subjects undergoing elective C-section. All subjects will remain in the hospital for up to 72 hours postsurgery.

Screening:

Subjects will be screened within 30 days prior to surgery; screening on the day of surgery will be allowed but is discouraged. During the screening visit, subjects will be assessed for any past or present medical conditions that in the opinion of the investigator would preclude them from study participation. After the informed consent form (ICF) is signed, a medical history, surgical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, alcohol breath test and urine drug screen, and clinical laboratory tests (hematology and chemistry) will be performed.

Day of Surgery:

Pre-operative medications: Use of pre-operative analgesics (eg, opioid medications, acetaminophen, nonsteroidal anti-inflammatory drugs [NSAIDs]) is prohibited.

Eligible subjects will be randomized in a blinded 1:1 ratio to either:

* Group 1: EXPAREL+bupivacaine TAP infiltration following spinal anesthesia
* Group 2: Active bupivacaine HCl TAP infiltration following spinal anesthesia On Day 1, prior to the C-section, all subjects will receive a intrathecal injection of 150 mcg preservative-free morphine for spinal injection (eg, Duramorph®) in conjunction with single-shot spinal anesthesia using 1.4-1.6 mL bupivacaine HCl 0.75% and 15 mcg fentanyl. If preservative-free morphine for spinal injection (eg, Duramorph) is unavailable because of a drug shortage, subjects may instead receive an intrathecal injection of 75 mcg preservative-free hydromorphone in conjunction with single-shot spinal anesthesia using 1.4-1.6 mL bupivacaine HCl 0.75% and 15 mcg fentanyl. A combined spinal epidural (CSE) anesthesia technique may also be used provided the epidural component is not used. Subjects who receive the epidural component of the CSE anesthesia must be immediately withdrawn from the study.

Intraoperative medications: The intraoperative use of the following medications is discouraged, but may be permitted if clinically indicated based on the investigator's discretion (all medications must be appropriately recorded [ie, drug, dose, and route of administration]): ketamine and midazolam (Versed®). Prophylactic use of dexamethasone for prevention of nausea and vomiting is prohibited.

After delivery of the baby and prior to the TAP infiltration, a small amount of lidocaine (<2 mL) may be administered subcutaneously to form a skin wheal over the area of the needle insertion site. A 2-point classic TAP block will be performed under ultrasound guidance within 1 hour (± 30 minutes) following skin incision closure of the C-section. A confirmatory ultrasound picture or video will be taken of each side of the abdomen after the TAP needle position has been established and following infiltration of study drug.

TAP infiltration: Subjects randomized to the EXPAREL+bupivacaine group (Group 1) will receive a single 20-mL dose of EXPAREL 266 mg expanded in volume with 20 mL normal saline plus 20 mL 0.25% bupivacaine for a total volume of 60 mL, administered as 30 mL (10 mL EXPAREL, 10 mL 0.25% bupivacaine HCl, and 10 mL saline) on each side of the abdomen. Subjects randomized to the active bupivacaine group (Group 2) will receive 20 mL 0.25% bupivacaine expanded in volume with 40 mL normal saline for a total volume of 60 mL, administered as 30 mL (10 mL 0.25% bupivacaine HCl and 20 mL saline) on each side of the abdomen.

Postsurgical Analgesia: Patient-controlled analgesia is not permitted. The following multimodal pain regimen will be initiated immediately following the delivery of the baby:

* IV ketorolac 15 mg once at the time of skin incision closure and prior to the TAP infiltration
* Intravenous (IV) acetaminophen 1000 mg at the time of skin incision closure
* Scheduled oral (PO) acetaminophen 650 mg beginning 6 hours from the administration of the single dose of IV acetaminophen at the end of surgery and then every 6 hours (q6h) for up to 72 hours or hospital discharge
* Scheduled PO ibuprofen 600 mg beginning 6 hours from the administration of the single dose of IV ketorolac at the end of surgery and then q6h for up to 72 hours or hospital discharge

The date, time, and dose of all standardized multimodal pain medications administered must be recorded. Note: The scheduled PO medication will be administered on a q6h schedule only through hospital discharge.

Rescue Medication: Subjects should only receive opioid rescue pain medication upon request for breakthrough pain. Postsurgical rescue medication will comprise PO immediate-release oxycodone (initiated at 5-10 mg every 4 hours [q4h] or as needed [PRN]). If a subject is unable to tolerate PO medication or fails the PO oxycodone rescue, IV morphine (initiated at 1-2 mg) or hydromorphone (initiated at 0.3-0.5 mg) may be administered q4h or PRN. All surgical and postsurgical opioid and other analgesics (pain medications) administered must be documented through Day 14 postsurgery. Additionally, an unscheduled pain intensity score using a 10-cm visual analog scale (VAS) must be completed immediately prior to any rescue medication while in the hospital.

Permitted medications for the prevention and treatment of possible medication side effects include the following and may be used at the discretion of the study site principal investigator:

* Ondansetron 4 mg IV immediately after delivery of the baby.
* Ondansetron 4 mg IV (should not exceed a maximum of 12 mg in a 24-hour period) for intraoperative and postoperative nausea and vomiting
* Metoclopramide 10 mg PO PRN for nausea and vomiting
* Nalbuphine IV 2.5 mg PRN for pruritus
* Naloxone IV 50-100 mcg PRN for pruritus.

Postsurgical Assessments:

Subjects will remain in the hospital for up to 72 hours postsurgery. Postsurgical assessments will include:

* Opioid use
* Time of first unassisted ambulation
* Pain intensity scores using a 10-cm VAS at rest
* Discharge readiness
* Subject's satisfaction with postsurgical pain control
* Overall benefit of anesthesia score (OBAS) questionnaire
* Quality of recovery 15-item questionnaire (QoR-15)

While in the hospital, subjects will be provided with a Patient Diary and will use the diary to record all scheduled and unscheduled VAS scores. For all scheduled assessments and unscheduled assessments in the hospital, subjects will assess, "How much pain are you experiencing right now" and a vertical mark will be placed on the VAS line to indicate the level of pain experienced at the time of assessment. If a subject is discharged prior to a scheduled VAS assessment, a member of the study site staff will contact the subject to remind her to complete the scheduled VAS assessment at the scheduled time and to record the assessment in the Patient Diary.

At hospital discharge, the subject will be instructed to record in the Patient Diary VAS pain intensity score daily and all pain medications taken following hospital discharge through Day 14.

At home, the subject will assess pain intensity at rest each day at noon (± 4 hours). This assessment should capture her average pain at rest in the prior 24 hours by assessing "What has been your average pain since your last pain assessment?" (ie, from noon on the previous day to the current assessment). At the same time, the subject should record any pain medication (medication name, date, time, and dose) taken in the prior 24 hours.

A phone call will be made to each subject on Day 14 for safety purposes and to inquire as to whether the subject has made any unscheduled phone calls or office visits related to pain; experienced any hospital readmission; or experienced an emergency room visit since hospital discharge. Adverse events (AEs) and serious adverse events (SAEs) will be recorded from the time the ICF is signed through Day 14.

ELIGIBILITY:
Inclusion Criteria:

1. Females 18 years of age and older at screening.
2. Term pregnancies of 37 to 42 weeks gestation, scheduled to undergo elective C-section.
3. American Society of Anesthesiology (ASA) physical status 1, 2, or 3.
4. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Subjects who, in the opinion of the study site principal investigator, have a high-risk pregnancy (eg, multiple gestations, pregnancy resulting from in vitro fertilization, gestational diabetes, end-term prolonged bed rest required for medical reasons).
2. Subjects with a pregnancy-induced medical condition or complication (eg, hypertension, pre-eclampsia, chorioamnionitis).
3. Subjects with 3 or more prior C-sections.
4. Pre-pregnancy body mass index >50 kg/m2 or otherwise not anatomically appropriate to undergo a TAP block.
5. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (eg, amide-type local anesthetics, opioids, bupivacaine, NSAIDs, spinal anesthesia).
6. Planned concurrent surgical procedure with the exception of salpingo-oophorectomy or tubal ligation.
7. Severely impaired renal or hepatic function (eg, serum creatinine level >2 mg/dL [176.8 μmol/L], blood urea nitrogen level >50 mg/dL [17.9 mmol/L], serum aspartate aminotransferase [AST] level >3 times the upper limit of normal [ULN], or serum alanine aminotransferase [ALT] level >3 times the ULN.)
8. Subjects at an increased risk for bleeding or a coagulation disorder (defined as platelet count less than 80,000 × 103/mm3 or international normalized ratio greater than 1.5)
9. Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the postsurgical period for pain that is not strictly related to the surgery and which may confound the postsurgical assessments.
10. Clinically significant medical disease in either the mother or baby that, in the opinion of the investigator, would make participation in a clinical study inappropriate. This includes any psychiatric or other disease in the mother that would constitute a contraindication to participation in the study or cause the mother to be unable to comply with the study requirements.
11. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
12. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study
13. Previous participation in an EXPAREL study. In addition, the subject will be ineligible to receive study drug and will be withdrawn from the study if she meets the following criteria during surgery:
14. Any clinically significant event or condition uncovered during the surgery (eg, excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postsurgical course.
15. Receives the epidural component of CSE anesthesia during participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for subjects undergoing elective Cesarean Section
Enrollment: 186 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Danesi, Study Director — Pacira Pharmaceuticals, Inc
Locations (12):
- United States (12):
  - Loma Linda University, Loma Linda, California
  - Stanford University Medical Center, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health Systems, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Peter's University Medical Center, New Brunswick, New Jersey
  - Columbia Universtiy Medical Center, New York, New York
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Inova Fairfax Medical Center, Falls Church, Virginia
  - West Virginia University School of Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nedeljkovic SS, Kett A, Vallejo MC, Horn JL, Carvalho B, Bao X, Cole NM, Renfro L, Gadsden JC, Song J, Yang J, Habib AS. Transversus Abdominis Plane Block With Liposomal Bupivacaine for Pain After Cesarean Delivery in a Multicenter, Randomized, Double-Blind, Controlled Trial. Anesth Analg. 2020 Dec;131(6):1830-1839. doi: 10.1213/ANE.0000000000005075. PMID 32739962

RESULTS

PARTICIPANT FLOW:
Groups:
- EXPAREL 266mg + Immediate Release (IR) Bupivacaine: 60 mL of a study drug mixture containing 20 mL EXPAREL (266 mg) combined with 20 mL bupivacaine HCl 0.25% (50 mg bupivacaine HCl or 44 mg bupivacaine HCl free base equivalents, calculated as 0.886 mg bupivacaine HCl free base = 1.0 mg bupivacaine HCl equivalents) and 20 mL normal saline (total mixture 60 mL) administered into the transversus abdominis plane (TAP), with half of the volume (30 mL) administered to each side of the abdomen.
- IR Bupivacaine: 60 mL of a study drug mixture containing 20 mL bupivacaine HCl 0.25% (50 mg) combined with 40 mL normal saline (total mixture 60 mL) administered into the TAP, with half of the volume (30 mL) administered to each side of the abdomen.
Period: Overall Study
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Started (Subject 263-0203 was randomized to bupivacaine HCl but received EXPAREL 266 mg. Subject 263-0203 is included in the IR bupivacaine group in this table.) | 96 | 90
Completed | 91 | 83
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Population: The safety analysis set includes all subjects who receive study drug. All analyses based on the safety set are by actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine | Total
Number analyzed (Participants) | 97 | 89 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (5.37) | 33.1 (4.43) | 33.4 (4.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 89 | 186
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 84 | 78 | 162
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 15 | 28
  White | 67 | 64 | 131
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 11 | 2 | 13
Region of Enrollment [Number; unit: participants]
  United States | 97 | 89 | 186
American Society of Anesthesiologists classification [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) classification was determined by physicians using the ASA Physical Status Classification System which assesses the patient's pre-anesthesia medical co-morbidities. ASA 1 patients would be considered a normal, healthy patient. ASA 2 is a patient with mild systemic disease (eg, smoker, well controlled diabetes or high blood pressure (HBP)). ASA 3 is a patient with severe systemic disease (eg poorly controlled diabetes or HBP). ASA 4 is a patient with severe systemic disease that is a constant threat to life (eg, recent myocardial infarction, stroke).
  Participants
    ASA 1 | 1 | 1 | 2
    ASA 2 | 90 | 80 | 170
    ASA 3 | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Postsurgical Opioid Consumption Through 72 Hours After TAP Infiltration During Elective Cesarean Section
Description: The primary endpoint is the total postsurgical opioid consumption (mg) in oral morphine equivalent dose (OMED) through 72 hours.
Time Frame: 0-72 hours
Population: Efficacy analysis set (also the modified intent-to-treat [mITT] analysis set) included all randomized subjects in the safety analysis set who underwent C-section and who also met the study criteria for correct TAP placement, local anesthetic dosing, and a multimodal post-operative analgesic regimen, with analysis based on randomized treatment (regardless of treatment received)
Measure: Least Squares Mean (Standard Error); unit: MED, mg
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Number analyzed (Participants) | 71 | 65
MED, mg | 15.5 (6.67) | 32.0 (6.25)
Statistical Analysis 1: Comparison: EXPAREL 266mg + Immediate Release (IR) Bupivacaine vs IR Bupivacaine; Test type: Superiority; p = 0.0117, ANCOVA; LSM treatment difference = -16.5, 95% CI 2-sided [-30.8 to -2.2]

2. Secondary Outcome: Area Under the Curve (AUC) for Visual Analog Scale (VAS) Pain Scores Through 72 Hours
Description: AUC for VAS pain scores through 72 hours. Pain intensity scores were measured on a 10-cm VAS (0 cm= "no pain" to 30 cm="pain as bad as it could be").
  Subjects were evaluated for pain intensity scores at rest using the 10-cm VAS at rest at 6, 12, 18, 24, 30, 36, 42, 48, and 72 hours after surgery and then once daily (at noon ± 4 hours) through Day 14. To assess pain intensity (VAS) at rest, the subject should rest quietly in a supine or seated position that does not exacerbate her postsurgical pain for 3-5 minutes before entering the pain score. While in the hospital, subjects are to assess, "How much pain are you experiencing right now?" and a vertical mark is placed on a 10-cm straight line to indicate the level of pain experienced at the time of assessment.
  Note higher AUC means more pain over time.
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm*hr
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Number analyzed (Participants) | 70 | 65
cm*hr | 147.9 (21.13) | 178.5 (19.78)
Statistical Analysis 1: Comparison: EXPAREL 266mg + Immediate Release (IR) Bupivacaine vs IR Bupivacaine; Test type: Non-Inferiority — Pre-specified non-inferiority margin of 36; p = 0.0020, ANCOVA; LSM treatment difference (SE) = -30.6, 95% CI 2-sided [-75.9 to 14.7]

3. Secondary Outcome: Opioid Spared Subjects Through 72 Hours
Description: Subjects were considered opioid-spared if:
  * For 0-72 hours opioid consumption, all doses add up to ≤15mg (oral morphine equivalent dose [OMED])
  * AND the overall benefit of anesthesia score (OBAS) score was 0 for questions 2, 3, 4, 5, and 6. For the OBAS questionnaire, 0 is considered minimal pain and 4 is considered maximum imaginable pain.
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Number analyzed (Participants) | 71 | 65
percent of participants | 53.5 | 24.7
Statistical Analysis 1: Comparison: EXPAREL 266mg + Immediate Release (IR) Bupivacaine; Test type: Superiority; p = 0.0012, LSM probability from logistic regression; Odds Ratio (OR) = 3.51, 95% CI 2-sided [1.557 to 7.906]

4. Secondary Outcome: Total Postsurgical Opioid Consumption Through 24 Hours
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: MED mg
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Number analyzed (Participants) | 71 | 65
MED mg | 2.4 (1.82) | 5.6 (1.70)
Statistical Analysis 1: Comparison: EXPAREL 266mg + Immediate Release (IR) Bupivacaine vs IR Bupivacaine; Test type: Superiority; p = .0543, ANCOVA; Least squares treatment difference = -3.2

5. Secondary Outcome: Total Postsurgical Opioid Consumption Through 48 Hours
Time Frame: 0-48 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: MED mg
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Number analyzed (Participants) | 71 | 65
MED mg | 9.1 (4.46) | 20.5 (4.18)
Statistical Analysis 1: Comparison: EXPAREL 266mg + Immediate Release (IR) Bupivacaine vs IR Bupivacaine; Test type: Superiority; p = .0096, ANCOVA; Least squares treatment difference = -11.4

6. Secondary Outcome: Total Postsurgical Opioid Consumption Through 168 Hours (Day 7)
Time Frame: 0-168 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: MED mg
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Number analyzed (Participants) | 71 | 65
MED mg | 23.3 (9.75) | 45.8 (9.13)
Statistical Analysis 1: Comparison: EXPAREL 266mg + Immediate Release (IR) Bupivacaine vs IR Bupivacaine; Test type: Superiority; p = .0175, ANCOVA; Least squares treatment difference = -22.4

7. Secondary Outcome: Total Postsurgical Opioid Consumption Through 336 Hours (Day 14)
Time Frame: 0-336 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: MED mg
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Number analyzed (Participants) | 71 | 65
MED mg | 28.2 (11.20) | 47.8 (10.49)
Statistical Analysis 1: Comparison: EXPAREL 266mg + Immediate Release (IR) Bupivacaine vs IR Bupivacaine; Test type: Superiority; p = .0542, ANCOVA; Least squares treatment difference = -19.6

8. Secondary Outcome: Time to First Rescue Medication Use
Description: The time to a subject's first use of an opioid medication for breakthrough pain after the end of surgery
Time Frame: From the end of surgery
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Number analyzed (Participants) | 71 | 65
hours | 53.2 [2.3 to 345.2] | 41.1 [2.5 to 345.7]
Statistical Analysis 1: Comparison: EXPAREL 266mg + Immediate Release (IR) Bupivacaine vs IR Bupivacaine; Test type: Superiority; p = 0.7536, Regression, Cox

9. Secondary Outcome: Opioid-Free Subjects Through 72 Hours
Description: Percentage of subjects who did not received an opioid rescue medication starting from the end of surgery through 72 hours
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Number; unit: percent of opioid-free participants
Arm/Group | EXPAREL 266mg + Immediate Release (IR) Bupivacaine | IR Bupivacaine
Number analyzed (Participants) | 71 | 65
percent of opioid-free participants | 51.9 | 48.6
Statistical Analysis 1: Comparison: EXPAREL 266mg + Immediate Release (IR) Bupivacaine vs IR Bupivacaine; Test type: Superiority; p = 0.3609, Regression, Logistic; Odds Ratio (OR) = 1.14

ADVERSE EVENTS:
Time Frame: Screening through postsurgical Day 14
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (eg, abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug without any judgment about causality.
  Serious AEs were defined as per clinicaltrials.gov.
Arm/Group | EXPAREL+Bupivacaine TAP Infiltration | Active Bupivacaine TAP Infiltration
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/89
Serious Adverse Events (participants affected / at risk) | 3/97 | 3/89
Other Adverse Events (participants affected / at risk) | 63/97 | 50/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL+Bupivacaine TAP Infiltration (N=97) | Active Bupivacaine TAP Infiltration (N=89)
Cardiomyopathy (Cardiac disorders) | 1 | 0
Abdominal wall hematoma (Gastrointestinal disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL+Bupivacaine TAP Infiltration (N=97) | Active Bupivacaine TAP Infiltration (N=89)
Constipation (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 24 | 11
Vomiting (Gastrointestinal disorders) | 12 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Dizziness (Nervous system disorders) | 6 | 5
Headache (Nervous system disorders) | 6 | 10
pruritis (Skin and subcutaneous tissue disorders) | 27 | 28
Rash (Skin and subcutaneous tissue disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication ≤18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for ≤120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Study Protocol (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT03176459/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT03176459/SAP_001.pdf